CLINICAL TRIAL: NCT02631707
Title: The Effect of High Protein Diets on Weight Loss and Lean Muscle Mass in Patients Awaiting Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Counties Manukau Health (Other)
Responsible Party: Principal Investigator, Andrew MacCormick, Investigator, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Highproteinbariatric
Record Dates: First submitted 2015-05-26; First posted 2015-12-16 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Diet, High-Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Standard Protein Diet (No Intervention): Control Arm Ministry of Health guidelines percentage energy from carbohydrate (50-55%), protein (10-15%) and fat (30%).
- Intervention High Protein Diet (Experimental): Intervention Arm Percentage energy from carbohydrate (40%), protein (30%) and fat (30%).
  Interventions: Other: High protein diet

INTERVENTIONS:
Other: High protein diet — The intervention diet is higher in protein than the control diet.
  Arms: Intervention High Protein Diet

SUMMARY:
All patients in CMDHB eligible for bariatric surgery are given a weight loss goal prior to surgery. It is unknown what the most effective diet is to lose weight, while still preserving muscle mass. The diet must also be acceptable and adhered to by patients. The aim of this study is to find out if a diet that is higher in protein and lower in carbohydrate than the standard Ministry of Health guidelines will have a greater effect on weight loss, preservation of lean muscle mass, surgical recovery score, adherence and acceptability.

DETAILED DESCRIPTION:
This pilot project is a randomised control trial with 24 participants. Diets will consist of 1200 and 1500kcals for females and males, respectively. The control arm is to receive the Ministry of Health guidelines percentage energy from carbohydrate (50-55%), protein (10-15%) and fat (30%). The intervention arm is to be lower in carbohydrate (40%), higher in protein (30%), moderate fat (30%). Participants will be required to continue the diet for at least 8 weeks while waiting for surgery. At baseline and at eight weeks their weight, hip circumference, waist circumference, neck circumference and body composition measurements will be taken. During their prescribed diet they are required to fill out a 3-day diet record. At the end of eight weeks the participants will perform a twenty-four hour urine collect for urea and creatinine. This will help determine adherence. Post-surgery (21-28 days) they will be required to complete a surgical recovery questionnaire and the above measurements will be recorded again. These data will be collected over a period beginning January 2015. It is expected that the intervention arm will have greater weight loss and better preservation of muscle mass leading to a better surgical recovery score. However because the intervention requires a higher intake of protein this may have an effect on adherence and acceptability in these participants. There are no known adverse effects of the intervention diet in the short term.

ELIGIBILITY:
Inclusion Criteria:

* Participants in this study will be patients eligible for bariatric surgery under CMDHB. These participants must have a BMI greater than 35kg/m2 with co-morbidities or a BMI greater than 40kg/m2.

Exclusion Criteria:

* Patients will be excluded from study if they do not attend surgeon or dietitian appointments. To be included in this study patients must be English speaking and weigh under 200kg.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Weight | After 8-weeks of diet and 21-28 days post bariatric surgery
  Scales
Change in Total body muscle mass | After 8-weeks of diet and 21-28 days post bariatric surgery
  Biometric scales

SECONDARY OUTCOMES:
Surgical recovery score | Surgical recovery score 21-28 days post surgery
  SRS tool
compliance | 8 weeks
  urinary creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D MacCormick, FRACS, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- Counties Manukau District Health Board, Auckland, New Zealand